CLINICAL TRIAL: NCT01316042
Title: A Double Blind Randomized Controlled 12 Month Trial of Metformin for the Treatment of Premature Pubarche in Girls
Brief Title: Metformin for the Treatment of Premature Pubarche in Girls
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment at collaborating sites
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35865
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-04

CONDITIONS: Premature Pubarche
Keywords: Puberty; Hormones
MeSH Terms: interventions — Sugars; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator): 2 pills per day for 12 months
  Interventions: Drug: sugar pill
- Metformin (Active Comparator): 2 212.5mg pill/day for 12 months
  Interventions: Drug: Metformin, glucophage

INTERVENTIONS:
Drug: sugar pill — 2 pills per day for 12 months
  Arms: sugar pill
Drug: Metformin, glucophage — 2 212.5mg pills/day for 12 months
  Other Names: metformin
  Arms: Metformin

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of metformin in lowering serum DHEAS levels in girls with premature pubarche and secondary, to observe changes in hormones associated with pubertal development including gonadotropins, sex steroids, insulin, adipocytokines, and growth factors.

ELIGIBILITY:
Inclusion Criteria:

1. Girls aged 4-10 with pubic hair prior to 8 years of age
2. Elevated DHEAS level above age normal levels
3. Informed consent from parents and assent from the girl

Exclusion Criteria:

1. Diagnosis of incomplete precocious puberty, peripheral precocious puberty, or evidence of any abnormal pituitary, hypothalamic, adrenal, thyroid, and gonadal function other than premature secretion of adrenal androgens.
2. Chronic illness requiring treatment that may interfere with growth and development, i.e. chronic steroid use, renal failure, etc.
3. 21-hydroxylase deficiency or other enzyme deficiency leading to the phenotype of congenital adrenal hyperplasia. 21-hydroxylase deficiency will be excluded in all patients by a fasting 17-hydroxyprogesterone (17-OHP) level < 2 ng/mL. In the case of elevated fasting 17-OHP levels, an ACTH stimulation test will be performed. A 1-hour stimulated value > 10 ng/mL will be an exclusion 82. As 21 hydroxylase deficiency is a congenital condition, any normal level in the past of 17-hydroxyprogesterone allows entry into this study.
4. Uncorrected thyroid disease (defined as TSH < 0.2 mIU/ML or > 5.5 mIU/mL). A normal level within the last year is adequate for entry.
5. Type I or Type II diabetes (defined as a fasting serum glucose > 125mg/dL on two occasions 83), or patients receiving anti-diabetic medications such as insulin, thiazolidinediones, acarbose, or sulfonylureas; patients currently receiving metformin XR for a diagnosis of Type I or Type II diabetes or for PCOS are also specifically excluded.
6. Liver disease defined as AST or ALT > 2 times normal or total bilirubin > 2.5 mg/dL.
7. Renal disease defined as BUN > 30 mg/dL or serum creatinine > 1.4 mg/dL.
8. Significant anemia (Hemoglobin < 10 mg/dL).
9. History of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident.
10. Known heart disease (New York Heart Association Class II or higher).
11. Enrolled simultaneously into other investigative studies that require medications, proscribe the study medications, or otherwise prevent compliance with the protocol. Patients who anticipate taking longer than a one month break during the protocol should not be enrolled.
12. Concomitant use other medications known to affect reproductive function or metabolism. These medications include growth hormone, IGF-1, medroxyprogesterone acetate, oral contraceptives, GnRH agonists and antagonists, anti-androgens, gonadotropins, anti-obesity drugs, somatostatin, diazoxide, ACE inhibitors, and calcium channel blockers. The washout period on all these medications will be three months.
13. Suspected adrenal or ovarian tumor secreting androgens or other ectopic steroid secreting tumor.
14. Suspected Cushing's syndrome.
15. Lactose intolerance (the placebo filler is lactose).
16. Known hypersensitivity to study medication, including ACTH and GnRH, or their excipients.
17. Any concomitant medical condition that in the opinion of the investigator, may expose a subject to unacceptable level of safety risk, or that affects subject compliance.
18. Subjects who anticipate having any surgery associated with restricted intake of fluids or radiological studies with contrast dye during the study period.
19. Any concomitant medical condition that in the opinion of the investigator, may expose a subject to unacceptable level of safety risk, or that affects subject compliance.

Ages: 4 Years to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Legro, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (3):
- United States (3):
  - Riley Hospital for Children, Indiana University School of Medicine, Indianapolis, Indiana
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh at the University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | Metformin
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Metformin | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 7.5 [6 to 9] | 6 [6 to 6] | 6.75 [6 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
DHEAS [Mean (Full Range); unit: ug/dL] | 177.0 [59.0 to 295.0] | 67.6 [51.0 to 84.2] | 122.3 [51.0 to 295.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum DHEAS Levels
Description: Change in DHEAS level was constructed per subject as the 1-year measurement minus the baseline measurement. Only descriptive statistics are provided, statistical tests were not conducted given the extremely small sample size per group.
Time Frame: 1 year
Measure: Mean (Full Range); unit: ug/dL
Arm/Group | Sugar Pill | Metformin
Number analyzed (Participants) | 2 | 1
ug/dL | 10.25 [-11.0 to 31.5] | 4.8 [4.8 to 4.8]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sugar Pill | Metformin
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=2) | Metformin (N=2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Pink eye (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study due to low recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No